CLINICAL TRIAL: NCT03704519
Title: A Phase I, Randomized, Placebo-controlled, Open-label, Three Period Crossover Study to Investigate the Effect of Darolutamide and Enzalutamide on Cerebral Blood Flow in Healthy Male Volunteers.
Brief Title: Imaging Study to Compare Effects of Darolutamide and Enzalutamide With Respect to Placebo on the Blood Flow in the Brain in Healthy Male Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 18426; 2018-001599-39 (EudraCT Number)
Record Dates: First submitted 2018-10-10; First posted 2018-10-12 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Cerebrovascular Circulation
Keywords: Healthy volunteers; Magnetic Resonance Imaging (MRI)
MeSH Terms: interventions — darolutamide; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Men_EPD (Experimental): Healthy male participants receive drugs in order Enzalutamide, Placebo and Darolutamide.
  Interventions: Drug: Darolutamide (BAY1841788); Drug: Enzalutamide; Other: Placebo
- Men_DEP (Experimental): Healthy male participants receive drugs in order Darolutamide, Enzalutamide and Placebo.
  Interventions: Drug: Darolutamide (BAY1841788); Drug: Enzalutamide; Other: Placebo
- Men_PDE (Experimental): Healthy male participants receive drugs in order Placebo, Darolutamide and Enzalutamide.
  Interventions: Drug: Darolutamide (BAY1841788); Drug: Enzalutamide; Other: Placebo
- Men_DPE (Experimental): Healthy male participants receive drugs in order Darolutamide, Placebo and Enzalutamide.
  Interventions: Drug: Darolutamide (BAY1841788); Drug: Enzalutamide; Other: Placebo
- Men_EDP (Experimental): Healthy male participants receive drugs in order Enzalutamide, Darolutamide and Placebo.
  Interventions: Drug: Darolutamide (BAY1841788); Drug: Enzalutamide; Other: Placebo
- Men_PED (Experimental): Healthy male participants receive drugs in order Placebo, Enzalutamide and Darolutamide.
  Interventions: Drug: Darolutamide (BAY1841788); Drug: Enzalutamide; Other: Placebo

INTERVENTIONS:
Drug: Darolutamide (BAY1841788) — 300 mg tablet darolutamide, once orally
  Other Names: Darolutamide: ODM-201
Drug: Enzalutamide — 4 x 40 mg capsules, once orally
  Other Names: MDV3100
Other: Placebo — 4 placebo tablets, once orally
  Other Names: Darolutamide-matching placebo

SUMMARY:
The current study would investigate the effects of a single dose of darolutamide and enzalutamide compared with placebo and compared to each other on human brain blood flow using arterial spin labeling magnetic resonance imaging (ASL-MRI), a non-invasive MRI technique. The change in cerebral blood flow was an indirect measure of brain penetration.

The risk of drug-associated CNS-related adverse events was likely to be correlated with the concentration of the drug in the brain. In contrast to enzalutamide, preclinical studies of darolutamide indicate that its brain penetration was much lower.

The aim of this study was to determine whether there was a difference between darolutamide and enzalutamide compared to placebo in cerebral blood flow and thus in brain penetration.

DETAILED DESCRIPTION:
The primary objective was to investigate drug-induced changes in grey matter cerebral blood flow during single-dose treatment with darolutamide or enzalutamide as compared to placebo using voxel-wise quantification of the grey matter for the entire brain.

The secondary objective was to investigate drug-induced changes in regional cerebral blood flow in brain areas related to cognitive function after single-dose treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are healthy as determined by medical history, physical examination, laboratory tests, and cardiac monitoring.

Exclusion Criteria:

* Existing or recent relevant diseases of vital organs (eg, liver diseases, heart diseases, renal disease, lung disease), central nervous system or other organs (eg, Diabetes mellitus, myasthenia gravis).
* Known contraindication to magnetic resonance imaging.
* Any structural variants or pathological abnormalities on structural brain MRI during screening.
* Any history of seizures including a febrile seizure in childhood, loss of consciousness, transient ischemic attack, or any condition that may pre-dispose to seizure.
* Participant with any type of neurological problems or history of psychiatric disorder, especially mood disorders including medical history with suicidal ideation and/or suicide attempts, which may disable the participant to consent to the study.
* Participants who use prescription or oral over the counter medications which might influence the study objectives, dietary/nutritional supplements, (including vitamins, natural and herbal remedies, eg, St. John's wort) within 2 weeks prior to first study intervention administration or during the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
Change in grey-matter cerebral blood flow of enzalutamide as compared to placebo | At 4 hours after drug
  Obtained by comparing whole brain grey matter quantitative voxel-by-voxel maps of cerebral blood flow/ perfusion (mL per 100g tissue per min) of enzalutamide to placebo. Measured in grey matter voxels with arterial spin labeling magnetic resonance imaging (ASL-MRI).
Change in grey-matter cerebral blood flow of darolutamide as compared to placebo | At 4 hours after drug
  Obtained by comparing whole brain grey matter quantitative voxel-by-voxel maps of cerebral blood flow/ perfusion (mL per 100g tissue per min) of darolutamide to placebo. Measured in grey matter voxels with ASL-MRI.
Change in grey-matter cerebral blood flow of enzalutamide as compared to darolutamide | At 4 hours after drug
  Obtained by comparing whole brain grey matter quantitative voxel-by-voxel maps of cerebral blood flow/ perfusion (mL per 100g tissue per min) of enzalutamide to darolutamide. Measured in grey matter voxels with ASL-MRI.

SECONDARY OUTCOMES:
Change in mean regional grey-matter cerebral blood flow in brain areas related to cognitive function during treatment of enzalutamide as compared to placebo | At 4 hours after drug
  Brain areas related to cognitive function comprise hippocampus and frontal cortex. Cerebral blood flow measured with ASL-MRI.
Change in mean regional grey-matter cerebral blood flow in brain areas related to cognitive function during treatment of darolutamide as compared to placebo | At 4 hours after drug
  Brain areas related to cognitive function comprise hippocampus and frontal cortex. Cerebral blood flow measured with ASL-MRI.
Change in mean regional grey-matter cerebral blood flow in brain areas related to cognitive function during treatment of enzalutamide as compared to darolutamide | At 4 hours after drug
  Brain areas related to cognitive function comprise hippocampus and frontal cortex. Cerebral blood flow measured with ASL-MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Centre for Neuroimaging Sciences, King's College, London, United Kingdom

REFERENCES:
- [Derived] Williams SCR, Mazibuko N, O'Daly O, Zurth C, Patrick F, Kappeler C, Kuss I, Cole PE. Comparison of Cerebral Blood Flow in Regions Relevant to Cognition After Enzalutamide, Darolutamide, and Placebo in Healthy Volunteers: A Randomized Crossover Trial. Target Oncol. 2023 May;18(3):403-413. doi: 10.1007/s11523-023-00959-5. Epub 2023 Apr 27. PMID 37103658
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/